CLINICAL TRIAL: NCT02735707
Title: Randomized, Embedded, Multifactorial Adaptive Platform Trial for Community- Acquired Pneumonia
Acronym: REMAP-CAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Australian and New Zealand Intensive Care Research Centre (Other); Medical Research Institute of New Zealand (Other); Unity Health (Other); Berry Consultants (Other); Global Coalition for Adaptive Research (Other); University of Pittsburgh Medical Center (Other); Intensive Care National Audit & Research Centre (Other); St. Marianna University School of Medicine (Other); Nat Intensive Care Surveillance - MORU (Other); National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Lennie Derde, Dr., UMC Utrecht
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1189-1653; 2015-002340-14 (EudraCT Number); 602525 (Other Grant/Funding Number: European Union, FP7-HEALTH-2013-INNOVATION-1, PREPARE); 16/631 (Other Grant/Funding Number: Health Research Council of New Zealand); APP1101719 (Other Grant/Funding Number: National Health and Medical Research Council, Australia); 158584 (Other Grant/Funding Number: Canadian Institute of Health Research); 2023-507889-89-00 (EU CTIS Number); 965313 (Other Grant/Funding Number: European Union, Horizon 2020 research and innovation programme, ECRAID-Base)
Record Dates: First submitted 2015-12-11; First posted 2016-04-13 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Community-acquired Pneumonia, Influenza, COVID-19
Keywords: Pneumonia; Lung Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Anti-Bacterial Agents; Moxifloxacin; Levofloxacin; Antibiotics; Hydrocortisone; Anti-Infective Agents; Ceftriaxone; Piperacillin-tazobactam; Ceftaroline; Amoxicillin-clavulanate; Oseltamivir; COVID-19; Influenza; Intensive care; Critical care; SARS-CoV-2; Vitamin C; Therapeutic Anticoagulation; Statin; Invasive Mechanical Ventilation; Convalescent plasma; Eritoran; Apremilast; DMX-200; Ivermectin; Baloxavir; Tocilizumab; Baricitinib; Imatinib
MeSH Terms: conditions — Community-Acquired Pneumonia; Influenza, Human; COVID-19; Pneumonia; Lung Diseases; Respiratory Tract Diseases; Respiratory Tract Infections | interventions — Ceftriaxone; Moxifloxacin; Levofloxacin; Piperacillin, Tazobactam Drug Combination; Ceftaroline; Amoxicillin-Potassium Clavulanate Combination; Hydrocortisone; Influenza Vaccines; Oseltamivir; Lopinavir; Hydroxychloroquine; Ritonavir; Ivermectin; Interferon beta-1a; Interleukin 1 Receptor Antagonist Protein; tocilizumab; sarilumab; Congresses as Topic; Ascorbic Acid; Aspirin; Clopidogrel; Prasugrel Hydrochloride; Ticagrelor; Simvastatin; eritoran; apremilast; Angiotensin-Converting Enzyme Inhibitors; Ramipril; Lisinopril; Perindopril; Enalapril; trandolapril; Captopril; Angiotensin Receptor Antagonists; Losartan; Valsartan; candesartan; Irbesartan; Telmisartan; olmesartan; Cysteamine; baloxavir; Imatinib Mesylate; baricitinib; nirmatrelvir and ritonavir drug combination; remdesivir; nirmatrelvir

STUDY DESIGN:
Intervention Model Description: Adaptive Bayesian Platform Trial evaluating multiple interventions in multiple domains
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (18):
- Antibiotic Domain (Other): Patients with community-acquired pneumonia admitted to participating intensive care units and requiring empiric antibiotic therapy will be randomised one of five antibiotic interventions.
  Note: the ceftaroline + macrolide intervention has been closed to recruitment.
  Interventions: Drug: Ceftriaxone; Drug: Moxifloxacin or Levofloxacin; Drug: Piperacillin-tazobactam; Drug: Ceftaroline; Drug: Amoxicillin-clavulanate
- Macrolide Duration Domain (Other): Patients with community-acquired pneumonia admitted to participating intensive care units who have been allocated to a beta-lactam antibiotic intervention in the Antibiotic Domain will be randomised to either a standard course or extended course of macrolide therapy
  Interventions: Drug: Standard course macrolide; Drug: Extended course macrolide
- Corticosteroid Domain (Other): Patients with community acquired pneumonia (CAP) admitted to participating hospitals will be randomised to a steroid use strategy.
  Note: this domain is now closed to patients with suspected or proven COVID-19. It remains open to patients with CAP without COVID-19.
  Note: the fixed-course hydrocortisone has been closed to recruitment
  Interventions: Other: No systemic corticosteroid; Drug: Fixed-duration Hydrocortisone; Drug: Shock-dependent hydrocortisone; Drug: Fixed-duration higher dose Hydrocortisone; Drug: Fixed-duration dexamethasone
- Influenza Antiviral Domain (Other): Patients with community-acquired pneumonia admitted to participating hospitals with microbiological testing confirmed influenza infection will be randomised to one of six interventions.
  Interventions: Other: No antiviral agent for influenza; Drug: Five-days oseltamivir; Drug: Ten-days oseltamivir; Drug: Baloxavir Marboxil; Drug: Five-days oseltamivir + baloxavir marboxil; Drug: Ten-days oseltamivir + baloxavir marboxil
- COVID-19 Antiviral Domain (Other): Patients admitted to participating hospitals with suspected or microbiological testing confirmed COVID-19 will be randomised to no ivermectin or ivermectin.
  Note: an earlier version of this domain evaluated lopinavir-ritonavir, hydroxychloroquine, and combination lopinavir-ritonavir and hydroxychloroquine against a 'no antiviral' control.
  This domain is now closed.
  Interventions: Other: No antiviral agent for COVID-19; Drug: Lopinavir / Ritonavir; Drug: Hydroxychloroquine; Drug: Hydroxychloroquine + lopinavir/ritonavir; Drug: Ivermectin
- COVID-19 Immune Modulation Domain (Other): Patients admitted to participating hospitals with suspected or microbiological testing confirmed COVID-19 will be randomised to one of up to five interventions.
  Note: this domain is now closed.
  Interventions: Other: No immune modulation for COVID-19; Drug: Interferon beta-1a; Drug: Anakinra; Drug: Tocilizumab; Drug: Sarilumab
- Anticoagulation Domain (Other): Patients admitted to participating intensive care units with suspected or microbiological testing confirmed COVID-19 will be randomised to an anticoagulation strategy.
  Note: A previous version of this domain evaluated local standard venous thromboprophylaxis against therapeutic dose anticoagulation. This domain is now closed.
  Interventions: Drug: Local standard venous thromboprophylaxis; Drug: Therapeutic dose anticoagulation; Drug: Conventional low dose thromboprophylaxis; Drug: Intermediate dose thromboprophylaxis; Drug: Continuation of therapeutic dose anticoagulation
- Immunoglobulin Domain (Other): Immunosuppressed patients admitted to participating hospitals with microbiological testing confirmed COVID-19 will be randomised to receive no immunoglobulin for COVID-19, or to receive high-titre convalescent plasma.
  Note: an earlier version of this domain was not restricted to immunosuppressed patients.
  Interventions: Other: No immunoglobulin; Biological: Convalescent plasma; Biological: Delayed administration of convalescent plasma
- Vitamin C Domain (Other): Patients admitted to participating hospitals with community-acquired pneumonia will be randomised to receive no vitamin C, or vitamin C.
  Note: this domain is now closed.
  Interventions: Other: No vitamin C; Drug: Vitamin C
- Simvastatin Domain (Other): Patients admitted to participating hospitals with suspected or microbiological testing confirmed COVID-19 will be randomised to receive no simvastatin, or simvastatin.
  Note: this domain is now closed.
  Interventions: Other: No simvastatin; Drug: Simvastatin
- Antiplatelet Domain (Other): Patients admitted to participating hospitals with suspected or microbiological testing confirmed COVID-19 will be randomised to receive no antiplatelet, aspirin, or site-preferred P2Y12 inhibitor.
  Note: this domain is now closed.
  Interventions: Other: No antiplatelet; Drug: Aspirin; Drug: P2Y12 inhibitor
- Mechanical Ventilation Domain (Other): Patients with community-acquired pneumonia admitted to participating intensive care units who are intubated and receiving invasive mechanical ventilation will be randomised to protocolised mechanical ventilation strategy, or clinician-preferred mechanical ventilation strategy
  Interventions: Procedure: Clinician-preferred mechanical ventilation strategy; Procedure: Protocolised mechanical ventilation strategy
- COVID-19 Immune Modulation (2) Domain (Other): Patients admitted to participating hospitals with microbiological testing confirmed COVID-19 will be randomised to receive one of three interventions.
  Note: this domain is now closed.
  Interventions: Other: No immune modulation for COVID-19; Drug: Eritoran; Drug: Apremilast
- ACE2 RAS Domain (Other): Patients admitted to participating hospitals with suspected or microbiological testing confirmed COVID-19 will be randomised to one of up to five renin-angiotensin system blockade strategies.
  Note: this domain is now closed.
  Interventions: Other: No renin-angiotensin system inhibitor; Drug: Angiotensin converting enzyme inhibitor; Drug: Angiotensin Receptor Blockers; Drug: ARB + DMX-200
- Cysteamine Domain (Other): Patients admitted to participating hospitals with severe community-acquired pneumonia, including patients with suspected or proven influenza or COVID-19, will be randomised to receive no cysteamine, or cysteamine.
  Note: this domain is now closed.
  Interventions: Other: No cysteamine; Drug: Cysteamine
- Endothelial Domain (Other): Patients admitted to participating hospitals with severe community-acquired pneumonia, including patients with suspected or proven influenza or COVID-19, will be randomised to receive no endothelial modulator or enteral imatinib.
  Interventions: Other: No endothelial modulator; Drug: Imatinib
- Influenza Immune Modulation (Other): Patients with community-acquired pneumonia admitted to participating intensive care units with microbiological testing confirmed influenza infection will be randomised to one of three interventions.
  Interventions: Other: No Immune Modulator for Influenza; Drug: Tocilizumab; Drug: Baricitinib
- COVID-19 Antiviral (II) Domain (Other): Patients admitted to participating hospitals with microbiological testing confirmed COVID-19 will be randomised to one of up to four interventions.
  Interventions: Other: No antiviral agent for COVID-19; Drug: Nirmatrelvir/ritonavir; Drug: Remdesivir; Drug: Nirmatrelvir/ritonavir + remdesivir

INTERVENTIONS:
Drug: Ceftriaxone — The duration and dose of empiric antibiotics will be determined by the treating clinician and local guidelines or practice.
  Arms: Antibiotic Domain
Drug: Moxifloxacin or Levofloxacin — The duration and dose of empiric antibiotics will be determined by the treating clinician and local guidelines or practice.
  Arms: Antibiotic Domain
Drug: Piperacillin-tazobactam — The duration and dose of empiric antibiotics will be determined by the treating clinician and local guidelines or practice.
  Arms: Antibiotic Domain
Drug: Ceftaroline — The duration and dose of empiric antibiotics will be determined by the treating clinician and local guidelines or practice.
  Note: this intervention is now closed.
  Arms: Antibiotic Domain
Drug: Amoxicillin-clavulanate — The duration and dose of empiric antibiotics will be determined by the treating clinician and local guidelines or practice.
  Arms: Antibiotic Domain
Drug: Standard course macrolide — Standard course of macrolide therapy, discontinued between study day 3 and the end of study day 5.
  The dosing of and route of administration is not protocolised, the following guidance is provided:
  * Initial IV administration of a macrolide is strongly preferred
  * The preferred IV macrolide is azithromycin, but IV clarithromycin may be substituted.
  * The preferred enteral macrolide is azithromycin, but enteral clarithromycin or roxithromycin may be substituted.
  Arms: Macrolide Duration Domain
Drug: Extended course macrolide — Extended course of macrolide therapy discontinued at the end of study day 14 or hospital discharge (whichever occurs first).
  The dosing of and route of administration is not protocolised, the following guidance is provided:
  * Initial IV administration of a macrolide is strongly preferred
  * The preferred IV macrolide is azithromycin, but IV clarithromycin may be substituted.
  * The preferred enteral macrolide is azithromycin, but enteral clarithromycin or roxithromycin may be substituted.
  Arms: Macrolide Duration Domain
Other: No systemic corticosteroid — Patients are not to receive any systemic corticosteroids, including hydrocortisone, to study day 28 or hospital discharge (whichever occurs first).
  Arms: Corticosteroid Domain
Drug: Fixed-duration Hydrocortisone — 50mg of intravenous hydrocortisone will be administered every 6 hours for up to 7 days.
  Note: this intervention is now closed.
  Arms: Corticosteroid Domain
Drug: Shock-dependent hydrocortisone — 50mg IV hydrocortisone every 6 hours while the patient is in septic shock
  Arms: Corticosteroid Domain
Drug: Fixed-duration higher dose Hydrocortisone — 100mg of intravenous hydrocortisone will be administered every 6 hours for up to 7 days.
  Note: this intervention was only available to patients with suspected or proven COVID-19 and is now closed.
  Arms: Corticosteroid Domain
Other: No antiviral agent for influenza — No antiviral agent intended to be active against influenza infection is to be administered
  Arms: Influenza Antiviral Domain
Drug: Five-days oseltamivir — Oseltamivir administered enterally twice daily for 5 days or until hospital discharge (whichever occurs first)
  Arms: Influenza Antiviral Domain
Drug: Ten-days oseltamivir — Oseltamivir administered enterally twice daily for 10 days or until hospital discharge (whichever occurs first)
  Arms: Influenza Antiviral Domain
Other: No antiviral agent for COVID-19 — No antiviral agent intended to be active against SARS-CoV-2 infection is to be administered
  Arms: COVID-19 Antiviral Domain
Drug: Lopinavir / Ritonavir — Lopinavir/ritonavir 400/100mg administered enterally, or 5ml 80/20mg per mL solution suspension via gastric tube, every 12 hours. Administered for a minimum of 5 days, including if discharged from ICU prior to end of study day 5. For patients discharged from ICU between study day 6 and study day 14, lopinavir/ritonavir is ceased at ICU discharge. Lopinavir/ritonavir is ceased at the end of study day 14 if the patient remains in ICU.
  Note: this intervention is now closed.
  Arms: COVID-19 Antiviral Domain
Drug: Hydroxychloroquine — Loading dose of 800mg hydroxychloroquine administered enterally every 6 hours until 2 doses have been administered. Subsequently, 400mg hydroxychloroquine will be administered enterally every 12 hours for 12 doses or ICU discharge (whichever occurs first).
  Note: this intervention is now closed.
  Arms: COVID-19 Antiviral Domain
Drug: Hydroxychloroquine + lopinavir/ritonavir — Lopinavir/ritonavir 400/100mg administered enterally, or 5ml 80/20mg per mL solution suspension via gastric tube, every 12 hours. Administered for a minimum of 5 days, including if discharged from ICU prior to end of study day 5. For patients discharged from ICU between study day 6 and study day 14, lopinavir/ritonavir is ceased at ICU discharge. Lopinavir/ritonavir is ceased at the end of study day 14 if the patient remains in ICU.
  Loading dose of 800mg hydroxychloroquine administered enterally every 6 hours until 2 doses have been administered. Subsequently, 400mg hydroxychloroquine will be administered enterally every 12 hours for 12 doses or ICU discharge (whichever occurs first).
  Note: this intervention is now closed.
  Arms: COVID-19 Antiviral Domain
Drug: Ivermectin — Ivermectin administered enterally at a dose of 0.2 mg/kg once daily with a maximum daily dose of 24mg/day.
  Note: this intervention is now closed.
  Arms: COVID-19 Antiviral Domain
Other: No immune modulation for COVID-19 — No immune modulating agent intended to be active against COVID-19 is to be administered.
  Note: this intervention is now closed.
  Arms: COVID-19 Immune Modulation (2) Domain; COVID-19 Immune Modulation Domain
Drug: Interferon beta-1a — IFN-β1a 10 μg will be administered as an intravenous bolus injection via a central or peripheral line. IFN-β1a will be administered once daily for 6 days or until ICU discharge, whichever occurs first.
  Note: this intervention is now closed.
  Other Names: IFN-β1a
  Arms: COVID-19 Immune Modulation Domain
Drug: Anakinra — A loading dose of 300mg anakinra will be administered as a bolus via central or peripheral line. This is followed by maintenance doses of 100mg of anakinra administered every 6 hours.
  In patients with renal impairment, anakinra will be administered on alternate days.
  Note: this intervention is now closed.
  Arms: COVID-19 Immune Modulation Domain
Drug: Tocilizumab — Tocilizumab will be administered as a single dose of 8mg/kg estimated or measured body weight, with a maximum total dose of 800mg.
  Tocilizumab will be administered as an IV infusion via central or peripheral line over a one-hour period.
  Note: this intervention is now closed.
  Arms: COVID-19 Immune Modulation Domain
Drug: Sarilumab — Sarilumab will be administered as a single dose of 400mg, via IV infusion through peripheral or central line over a one-hour period.
  Note: this intervention is now closed.
  Arms: COVID-19 Immune Modulation Domain
Drug: Local standard venous thromboprophylaxis — Standard venous thromboprophylaxis that complies with local guidelines or usual practice will be administered for 14 days following randomisation or until hospital discharge, whichever occurs first.
  Note: this intervention is now closed.
  Arms: Anticoagulation Domain
Drug: Therapeutic dose anticoagulation — Patients will be administered either low molecular weight heparin (LMWH) or unfractionated heparin (UFH) to achieve systemic anticoagulation. Either agent may be used and the same patient may be switched between UFH and LMWH at the discretion of the treating clinician.
  Note: this intervention is now closed.
  Arms: Anticoagulation Domain
Drug: Conventional low dose thromboprophylaxis — Low dose thromboprophylaxis will be administered for 14 days following randomisation or until hospital discharge, whichever occurs first. Dosing is outlined in the relevant protocol documents for this domain.
  Arms: Anticoagulation Domain
Drug: Intermediate dose thromboprophylaxis — Intermediate dose thromboprophylaxis will be administered for 14 days following randomisation or until hospital discharge, whichever occurs first. Dosing is outlined in the relevant protocol documents for this domain.
  Arms: Anticoagulation Domain
Drug: Continuation of therapeutic dose anticoagulation — Patients already receiving therapeutic dose anticoagulation at the time of randomisation to this intervention will be administered either unfractionated heparin by IV infusion or low-molecular weight heparin to achieve systemic anticoagulation according to local practice for acute VTE treatment for 14 days following randomisation or until hospital discharge, whichever occurs first.
  Note: this intervention is now closed.
  Arms: Anticoagulation Domain
Other: No immunoglobulin — No immunoglobulin intended to be active against SARS-CoV-2 infection is to be administered.
  Arms: Immunoglobulin Domain
Biological: Convalescent plasma — Patients will receive at least one and no more than two units of ABO compatible convalescent plasma within 48 hours of randomisation.
  Arms: Immunoglobulin Domain
Biological: Delayed administration of convalescent plasma — Note: this intervention is now closed.
  Arms: Immunoglobulin Domain
Other: No vitamin C — No high dose intravenous vitamin C is to be administered
  Note: this intervention is now closed.
  Arms: Vitamin C Domain
Drug: Vitamin C — Intravenous Vitamin C 50mg/kg administered every 6 hours for 16 doses
  Note: this intervention is now closed.
  Arms: Vitamin C Domain
Other: No antiplatelet — No antiplatelet agent or NSAID to be administered.
  Note: this intervention is now closed.
  Arms: Antiplatelet Domain
Drug: Aspirin — Aspirin administered at either 75mg or 100mg once per day for 14 days or until hospital discharge, whichever occurs first.
  Note: this intervention is now closed.
  Other Names: acetylsalicylic acid
  Arms: Antiplatelet Domain
Drug: P2Y12 inhibitor — Site-selected P2Y12 inhibitor:
  * Clopidogrel: administered 75 mg once per day for 14 days or until hospital discharge, whichever occurs first.
  * Prasugrel: If patient is aged less than 75 years and measured or estimated weight if 60kg or more, and initial loading dose of prasugrel 60 mg will be administered, followed by maintenance dose of 10 mg per day.
  * Ticagrelor: administered enterally at 60mg twice daily for 14 days or until hospital discharge, whichever occurs first.
  Note: this intervention is now closed.
  Other Names: Clopidogrel; Prasugrel; Ticagrelor
  Arms: Antiplatelet Domain
Other: No simvastatin — No simvastatin intended to be active against COVID-19 is to be administered
  Note: this intervention is now closed.
  Arms: Simvastatin Domain
Drug: Simvastatin — Simvastatin 80mg administered once daily via enteral route, while the patient remains in hospital up to 28 days after randomisation
  Note: this intervention is now closed.
  Arms: Simvastatin Domain
Drug: Eritoran — Eritoran initiated with a 26.24 mg loading dose (6.56 mg/h IV for 4 hours), followed by a second 13.12 mg loading dose (6.56 mg/h IV for 2 hours) at 12 hours after initiation. Patients will then receive twenty-six 6.56 mg maintenance doses (3.28 mg/h IV for 2 hours) every 12 hours thereafter (total of 14 days). Dosing will be stopped if the patient is discharged from hospital
  Note: this intervention is now closed.
  Arms: COVID-19 Immune Modulation (2) Domain
Drug: Apremilast — Apremilast administered 30mg twice daily for 14 days or until hospital discharge, whichever occurs first.
  Note: this intervention is now closed.
  Arms: COVID-19 Immune Modulation (2) Domain
Procedure: Clinician-preferred mechanical ventilation strategy — Clinician-preferred ventilation strategy, including mode of ventilation and all ventilatory parameters
  Arms: Mechanical Ventilation Domain
Procedure: Protocolised mechanical ventilation strategy — Invasive mechanical ventilation strategy delivered as outlined in relevant protocol documents for this domain.
  Arms: Mechanical Ventilation Domain
Other: No renin-angiotensin system inhibitor — No RAS inhibitor (i.e. no ACEi or ARB) is to be administered up to the end of study day 10.
  Note: this intervention is now closed.
  Arms: ACE2 RAS Domain
Drug: Angiotensin converting enzyme inhibitor — Site-preferred ACEi agent administered as directed by the treating clinician for 10 days or until hospital discharge, whichever occurs first.
  Note: this intervention is now closed.
  Other Names: Ramipril; Lisinopril; Perindopril; Enalapril; Trandolapril; Captopril
  Arms: ACE2 RAS Domain
Drug: Angiotensin Receptor Blockers — Site-preferred ARB agent administered as directed by the treating clinician for 10 days or until hospital discharge, whichever occurs first.
  Note: this intervention is now closed.
  Other Names: Losartan; Valsartan; Candesartan; Irbesartan; Telmisartan; Olmesartan
  Arms: ACE2 RAS Domain
Drug: ARB + DMX-200 — Site-preferred ARB agent administered in combination with DMX-200 for 10 days or until hospital discharge, whichever occurs first.
  ARB administered as directed by the treating clinician. DMX-200 administered enterally at a dose of 120mg twice daily.
  Note: this intervention is now closed.
  Arms: ACE2 RAS Domain
Other: No cysteamine — No cysteamine to be administered until the end of study day 10 or hospital discharge, whichever occurs first.
  Note: this intervention is now closed.
  Arms: Cysteamine Domain
Drug: Cysteamine — Cysteamine administered every 8 hours at a dose of 5 mg/kg estimated or measured body weight (maximum dose of 500mg), for ten days or until ICU discharge, whichever occurs first.
  Note: this intervention is now closed.
  Arms: Cysteamine Domain
Drug: Fixed-duration dexamethasone — 6 mg of IV or enteral dexamethasone will be administered daily for up to 10 days while in hospital.
  Arms: Corticosteroid Domain
Drug: Baloxavir Marboxil — Baloxavir marboxil administered on days 1 and 4 post-randomisation.
  Arms: Influenza Antiviral Domain
Drug: Five-days oseltamivir + baloxavir marboxil — Oseltamivir administered enterally twice daily for 5 days or until hospital discharge (whichever occurs first), in addition to baloxavir marboxil administered on days 1 and 4 post-randomisation.
  Arms: Influenza Antiviral Domain
Drug: Ten-days oseltamivir + baloxavir marboxil — Oseltamivir administered enterally twice daily for 10 days or until hospital discharge (whichever occurs first), in addition to baloxavir marboxil administered on days 1 and 4 post-randomisation.
  Arms: Influenza Antiviral Domain
Other: No endothelial modulator — No endothelial modulator (imatinib or another tyrosine kinase inhibitor targeting the same pathway as imatinib) is to be administered.
  Arms: Endothelial Domain
Drug: Imatinib — Enteral imatinib will be administered as a single 800mg loading dose (study day 1) followed by 400mg daily until study day 14 or discharge.
  Arms: Endothelial Domain
Other: No Immune Modulator for Influenza — No immune modulating agent intended to be active against influenza is to be administered.
  Arms: Influenza Immune Modulation
Drug: Tocilizumab — Tocilizumab will be administered as a single dose of 8mg/kg estimated or measured body weight, with a maximum total dose of 800mg. In children weighing less than 30kg, tocilizumab dose will be 12mg/kg.
  Tocilizumab will be administered as an IV infusion via central or peripheral line over a one-hour period.
  Arms: Influenza Immune Modulation
Drug: Baricitinib — Baricitinib will be administered at a dose that is determined by age and renal function, for up to 10 days or hospital discharge (whichever occurs first).
  Arms: Influenza Immune Modulation
Other: No antiviral agent for COVID-19 — No antiviral agent intended to be active against SARS-CoV-2 infection is to be administered
  Arms: COVID-19 Antiviral (II) Domain
Drug: Nirmatrelvir/ritonavir — Nirmatrelvir-ritonavir will be administered at a dose that is dependent on renal function, for five days.
  Other Names: Paxlovid
  Arms: COVID-19 Antiviral (II) Domain
Drug: Remdesivir — Remdesivir is administered at 200 mg on day one followed by 100 mg daily for a further four doses (i.e., for five doses in total) or until hospital discharge, whichever occurs first.
  Arms: COVID-19 Antiviral (II) Domain
Drug: Nirmatrelvir/ritonavir + remdesivir — Nirmatrelvir-ritonavir will be administered at a dose that is dependent on renal function, for five days. Remdesivir is administered at 200 mg on day one followed by 100 mg daily for a further four doses (i.e., for five doses in total) or until hospital discharge, whichever occurs first.
  Arms: COVID-19 Antiviral (II) Domain

SUMMARY:
REMAP-CAP is a randomised, embedded, multifactorial, adaptive platform trial for community-acquired pneumonia.

The purpose of this study is to evaluate the effect of a range of interventions to improve outcome of patients admitted to intensive care with community-acquired pneumonia.

In addition, REMAP-CAP provides and adaptive research platform for evaluation of multiple treatment modalities in the event of a respiratory pandemic such as COVID-19.

REMAP-COVID is a sub-platform of REMAP-CAP that evaluates treatments specific to COVID-19 in the United States of America.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) that is of sufficient severity to require admission to an intensive care unit (ICU) is associated with substantial mortality.

Patients with pneumonia who are being treated in an ICU will receive therapy that consists of many different treatments, as many as 20 or 30. These treatments act together to treat both the infection and its effects on the body. When treating a patient, doctors choose from many different treatments, most of which are known or believed to be safe and effective. However, doctors don't always know which treatment option is the better one, as individuals or groups of individuals may respond differently. This study aims to help doctors understand which treatments work best.

This clinical study has been designed in a way that allows the information from patients already in the study to help new patients joining the study. Most studies aren't able to do that. REMAP-CAP has been designed to:

* Evaluate multiple treatment strategies, at the same time, in the same patient.
* Reach platform conclusions when sufficient data is accrued, rather than when a pre-specified sample size is reached
* Utilise data that is already accrued to increase the likelihood that patients within the trial are randomised to treatments that are more likely to be beneficial
* New questions can be substituted into the trial as initial questions are answered, meaning that the trial can be perpetual or open-ended
* Interactions between interventions in different domains can be evaluated

It is reasonable to presume that any pandemic respiratory infection of major significance to public health will manifest as life-threatening respiratory infection including Severe Acute Respiratory illness and severe Community Acquired Pneumonia (CAP) with concomitant admission to hospital, and for some patients, admission to an Intensive Care Unit (ICU). Previous pandemics and more localized outbreaks of respiratory emerging infections have resulted in severe CAP and ICU admission.

Previous pandemics and outbreaks of emerging infectious diseases have outlined the urgent need for evidence, preferably from Randomized Controlled Trials (RCTs), to guide best treatment. However, there are substantial challenges associated with being able to organize such trials when the time of onset of a pandemic and its exact nature are unpredictable. As an adaptive platform trial that enrolls patients during the interpandemic period, REMAP-CAP is ideally positioned to adapt, in the event of a respiratory pandemic, to evaluate existing treatments as well as novel approaches.

ELIGIBILITY:
REMAP-CAP PLATFORM INCLUSION CRITERIA:

1. Adult patient admitted to an ICU for severe CAP within 48 hours of hospital admission with:

   1. symptoms or signs or both that are consistent with lower respiratory tract infection AND
   2. Radiological evidence of new onset consolidation (in patients with pre-existing radiological changes, evidence of new infiltrate)
2. Up to 48 hours after ICU admission, receiving organ support with one or more of:

   1. Non-invasive or Invasive ventilatory support;
   2. Receiving infusion of vasopressor or inotropes or both

PLATFORM EXCLUSION CRITERIA:

1. Healthcare-associated pneumonia:

   1. Prior to this illness, is known to have been an inpatient in any healthcare facility within the last 30 days
   2. Resident of a nursing home or long term care facility
2. Death is deemed to be imminent and inevitable during the next 24 hours AND one or more of the patient, substitute decision maker or attending physician are not committed to full active treatment
3. Previous participation in this REMAP within the last 90 days

REMAP-COVID PLATFORM INCLUSION CRITERIA

1. Adult patients (≥ 18 years) admitted to hospital with acute illness due to suspected or proven pandemic infection.

REMAP-COVID PLATFORM EXCLUSION CRITERIA

1. Death is deemed to be imminent and inevitable during the next 24 hours AND one or more of the patient, substitute decision maker or attending physician are not committed to full active treatment
2. Patient is expected to be discharged from hospital today or tomorrow
3. More than 14 days have elapsed while admitted to hospital with symptoms of an acute illness due to suspected or proven pandemic infection.
4. Previous participation in this REMAP within the last 90 days

DOMAIN-SPECIFIC ELIGIBLE CRITERIA:

Each domain may have additional eligibility criteria. Refer to the study website for more information (www.remapcap.org).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2016-04-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Day 90
Days alive and not receiving organ support in ICU | Day 21
  Primary end-point for patients with suspected or proven COVID-19 pandemic infection

SECONDARY OUTCOMES:
ICU Mortality | Day 90
ICU length of stay | Day 90
Hospital length of stay | Day 90
Ventilator free days | Day 28
Organ failure free days | Day 28
All-cause mortality | 6 months
Health-related Quality of life assessment | 6 months
  EQ5D-5L and WHODAS 2.0 (not completed in all regions)
Proportion of intubated patients who receive a tracheostomy | Day 28
Destination at time of hospital discharge | Free text Day 90
  Characterised as home, rehabilitation hospital, nursing home or long-term care facility, or another acute hospital
Readmission to the index ICU during the index hospitalization | Day 90
World Health Organisation 8-point ordinal scale outcome | Hospital discharge

OTHER OUTCOMES:
Occurrence of multi-resistant organism colonisation/infection | Day 90, censored at hospital discharge
  Antibiotic Domain specific outcome
Occurrence clostridium difficile | Day 90, censored at hospital discharge
  Antibiotic Domain specific outcome
Occurrence of serious ventricular arrhythmia (including ventricular fibrillation) or sudden unexpected death | Day 90, censored at hospital discharge
  Macrolide Duration Domain specific outcome.
Change from baseline influenza virus levels in upper and lower respiratory tract specimens | Day 3, up to Day 7
  Antiviral Domain specific outcome. Only required at selected sites.
Confirmed deep vein thrombosis | Between randomisation and hospital discharge
  Domain-specific outcome for Anticoagulation, Immunoglobulin, and Antiplatelet Domains.
Confirmed pulmonary embolism | Between randomisation and hospital discharge
  Domain-specific outcome for Anticoagulation, Immunoglobulin, and Antiplatelet Domains.
Confirmed ischaemic cerebrovascular event | Between randomisation and hospital discharge
  Domain-specific outcome for Anticoagulation, Immunoglobulin, and Antiplatelet Domains.
Total red blood cell units transfused | Between randomisation and end of study day 15
  Domain-specific outcome for Anticoagulation and Antiplatelet Domains.
Confirmed acute myocardial infarction | Between randomisation and hospital discharge
  Domain-specific outcome for Anticoagulation, Immunoglobulin, and Antiplatelet Domains.
Peak troponin | Between randomisation and end of study day 15
  Domain-specific outcome for Anticoagulation and Antiplatelet Domains.
Major bleeding event | Between randomisation and end of study day 15
  Domain-specific outcome for Anticoagulation and Antiplatelet Domains.
Other confirmed thrombotic event, including mesenteric ischaemia and limb ischaemia | Between randomisation and hospital discharge
  Domain-specific outcome for Anticoagulation, Immunoglobulin, and Antiplatelet Domains.
Acute kidney injury (KDIGO stage >= 2 acute kidney injury) | Between randomisation and 7 days
  Domain-specific outcome for ACE2 RAS Domain
Change from baseline to peak creatinine | Between randomisation and 14 days
  Domain-specific outcome for ACE2 RAS Domain
Angioedema | Between randomisation and end of study day 12
  Domain-specific outcome for ACE2 RAS Domain
Change from baseline AST, ALT and bilirubin | Between randomisation and 14 days
  Domain-specific outcome for ACE2 RAS Domain

CONTACTS AND LOCATIONS:
Overall Officials: Steve Webb, Prof, Study Chair — Monash University, Study Chair REMAP-CAP Australia; Colin McArthur, Dr, Study Chair — Medical Research Institute of New Zealand, Study Chair REMAP-CAP New Zealand; Marc Bonten, Prof, Study Chair — UMC Utrecht, Study Chair REMAP-CAP Europe; Lennie Derde, MD, Study Chair — UMC Utrecht, Coordinating Investigator REMAP-CAP Europe; John Marshall, Prof, Study Chair — Unity Health Toronto, Study Chair REMAP-CAP Canada; Derek Angus, Prof, Study Chair — University of Pittsburgh Medical Center, Study Chair REMAP-CAP USA
Locations (408):
- United States (11):
  - University of Florida, Jacksonville, Florida
  - Augusta University, Augusta, Georgia
  - University of Illinois Health, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Centre, Pittsburgh, Pennsylvania
  - Brown University - Rhode Island Hospital, Providence, Rhode Island
- Australia (59):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Blacktown Hospital, Blacktown, New South Wales
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Sutherland Hospital, Caringbah, New South Wales
  - Concord Hospital, Concord, New South Wales
  - Dubbo Base Hospital, Dubbo, New South Wales
  - Northern Beaches Hospital, Frenchs Forest, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Orange Health Service, Orange, New South Wales
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Wollongong Hospital, Sydney, New South Wales
  - Wagga Wagga Base Hospital, Wagga Wagga, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Darwin Hospital,, Darwin, Northern Territory
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - The Prince Charles Hospital, Brisbane, Queensland
  - Mater Hospital Brisbane, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Caboolture Hospital, Caboolture, Queensland
  - Queen Elizabeth II Jubilee Hospital, Coopers Plains, Queensland
  - Logan Hospital, Logan City, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Launceston Hospital, Launceston, Tasmania
  - Ballarat Base Hospital, Ballarat, Victoria
  - Bendigo Hospital, Bendigo, Victoria
  - Casey Hospital, Berwick, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - Angliss Hospital, Ferntree Gully, Victoria
  - Footscray Hospital, Footscray, Victoria
  - University Hosptial Geelong, Geelong, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
  - Maroondah Hospital, Ringwood East, Victoria
  - Sunshine Hospital, Sunshine, Victoria
  - Werribee Mercy Hospital, Werribee, Victoria
  - St John of God Hospital Midland, Midland, Western Australia
  - St John of God Hospital Murdoch, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
  - St John of God Subiaco, Subiaco, Western Australia
- Belgium (3):
  - CHU de Charleroi - Hôpital Civil Marie Curie, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - CHU Namur site Godinne, Namur
- Canada (40):
  - Foothills Medical Centre, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Royal Alexandra Hospital, Alberta, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Surrey Memorial Hospital, Surrey, British Columbia
  - St Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Grace Hospital, Winnipeg, Manitoba
  - Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - The Moncton Hospital, Fredericton, New Brunswick
  - The Saint John General Hospital, Fredericton, New Brunswick
  - William Osler Health System, Brampton, Ontario
  - Brantford General Hospital, Brantford, Ontario
  - Hamilton general Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - St Mary's General Hospital, Kitchener, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health, Saint Catharines, Ontario
  - Thunder Bay General Hospital, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital Unity Health Toronto, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - St Joseph's Health Centre, Toronto, Ontario
  - CIUSS Chaudieres-Appalaches (Levis), Lévis, Quebec
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
  - Hôpital Fleury, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - IUCPQ-UL, Québec, Quebec
  - Centre Hospitalier de l'Université de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Saskatoon, Saskatchewan
- Universidad de La Sabana, Chía, Cundinamarca, Colombia
- Croatia (3):
  - General County Hospital Požega, Požega
  - University Hospital Centre Zagreb, Zagreb
  - University Hospital for Infectious Diseases, Zagreb
- Czechia (2):
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Teplice Hospital, Teplice
- Tartu University Hospital, Tartu, Estonia
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
- France (24):
  - CH Argenteuil, Argenteuil
  - Centre Hospitalier Henri Mondor d'Aurillac, Aurillac
  - Beauvais General Hospital, Beauvais
  - Hopital Nord Franche-Comte, Belfort
  - Centre hospitalier Bethune Beuvry, Béthune
  - Ambroise Pare Hospital, Boulogne-Billancourt
  - CH de Dax, Dax
  - Centre Hospitalier de Dieppe, Dieppe
  - CHU Dijon Bourgogne, Dijon
  - Hopital Simone Veil Eaubonne, Eaubonne
  - Sud Essonne Hospital Etampes, Étampes
  - Hospital Raymond Poincare, Garches
  - CHD Vendee, La Roche-sur-Yon
  - Centre Hospitalier Le Mans, Le Mans
  - CHU Dupuytren, Limoges
  - Centre Hospitalier de Melun, Melun
  - Centre Hospitalier Layne - Mont-de-Marsan, Mont-de-Marsan
  - Centre Hospitalier des Pays de Morlaix, Morlaix
  - CHR d'Orleans, Orléans
  - Lariboisiere Hospital, Paris
  - Hopital Tenon, Paris
  - Nouvel Hopital Civil Strasbourg, Strasbourg
  - Hopital de Hautepierre Strasbourg, Strasbourg
  - CHRU Tours Hopital Bretonneau, Tours
- Germany (17):
  - Charité - Universitätsmedizin Berlin - Infektiologie und Pneumologie, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Charite Universitätsmedizin Berlin, Berlin
  - Vivantes Humboldt-Klinikum, Berlin
  - University Hospital of Cologne, Cologne
  - Carl-Thiem-Klinikum Cottbus, Cottbus
  - Klinikum Dortmund, Dortmund
  - Elisabeth Hospital Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - University Medical Center Hamburg-Eppendorf (UKE), Hamburg
  - Universitätsklinikum Jena, Jena
  - University Hospital Leipzig, Leipzig
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar der TU München, München
  - Universitätsklinikum Münster, Münster
  - Universitäts Klinikum Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (2):
  - Jósa András County Hospital, Nyíregyháza
  - Almási Balogh Pál Kórház, Ózd
- India (4):
  - Apollo Main Hospital, Chennai, Tamil Nadu
  - Apollo First Med Hospital, Chennai, Tamil Nadu
  - Apollo Vanagaram Hospital, Chennai, Tamil Nadu
  - Apollo Speciality Hospital - OMR, Chennai, Tamil Nadu
- Ireland (5):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Waterford, Waterford
- Israel (3):
  - Rambam Medical Center, Haifa
  - Beilinson Hospital, Rabin Medical Center, Petah Tikva
  - The Baruch Padeh Medical Center, Poria – Neve Oved
- Italy (8):
  - AO Spedali Civili di Brescia, Brescia
  - Humanitas Research Hospital, Milan
  - Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Istituto Mediterraneo per i Trapianti e Terapie ad alta specializzazione, Palermo
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale Infermi di Rimini, Rimini
- Japan (10):
  - St Marianna University School of Medicine, Kawasaki, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - St. Marianna University Yokohama City Seibu Hospital, Yokohama, Kanagawa
  - Saiseikai Kumamoto Hospital, Minami, Kumamoto
  - Osaka City General Hospital, Osaka
  - Nerima Hikarigaoka Hospital, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Tokyo
  - Itabashi Chuo Medical Center, Tokyo
  - Tokyo bay Urayasu-Ichikawa Medical Center, Tokyo
  - Wakayama Medical University, Wakayama
- Nepal (4):
  - Chitwan Medical College, Bharatpur
  - Grande International Hospital, Kathmandu
  - Hospital for Advanced Medicine and Surgery (HAMS), Kathmandu
  - Nepal Mediciti, Kathmandu
- Netherlands (19):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - ZGT Almelo, Almelo
  - Meander Medisch Centrum, Amersfoort
  - OLVG, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Deventer Hospital, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Maxima Medisch Centrum Eindhoven, Eindhoven
  - Martini Hospital Groningen, Groningen
  - University Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud University Medical Center, Nijmegen
  - Laurentius Hospital, Roermond
  - Maasstad Ziekenhuis, Rotterdam
  - Hagaziekenhuis, The Hague
  - Bernhoven Hospital, Uden
  - University Medical Center Utrecht, Utrecht
- New Zealand (11):
  - North Shore Hospital, Auckland
  - CVICU, Auckland City Hospital, Auckland
  - DCCM, Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Taranaki Base Hospital, New Plymouth
  - Rotorua Hospital, Rotorua
  - Tauranga Hospital, Tauranga
  - Wellington Regional Hospital, Wellington
  - Whangarei Hospital, Whangarei
- Pakistan (5):
  - Ziauddin University Hospital Clifton Campus, Karachi, Sindh
  - Abbasi Shaheed Hospital, Karachi, Sindh
  - National Institute of Cardiovascular Diseases, Karachi, Karachi, Sindh
  - South City Hospital, Karachi, Karachi, Sindh
  - Ziauddin University North Nazimabad Campus, Karachi, Sindh
- Portugal (3):
  - Centro Hospitalar do Medio Tejo, Abrantes
  - Hospital Ocidental, Lisbon
  - Hospital Lusíadas Lisbon, Lisbon
- Clinical Hospital of Infectious and Tropical Diseases "Dr. Victor Babes", Bucharest, Romania
- King Abdulaziz Medical City, Riyadh, Saudi Arabia
- Serbia (3):
  - University Clinical Centre of Serbia, Belgrade
  - University Hospital Center Dr Dragiša Mišović, Belgrade
  - Clinical Centre of Niš, Niš
- Slovenia (2):
  - University Clinic of Respiratory and Allergic Diseases Golnik, Golnik
  - University Medical Centre Maribor, Maribor
- Spain (10):
  - Hospital del Mar, Barcelona
  - Hospital Universitario de Jerez, Cadiz
  - Reina Sofia University Hospital, Córdoba
  - Ramon y Cajal University Hospital, Madrid
  - Hospital Regional de Málaga, Málaga
  - Hospital Universitario de Ourense, Ourense
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Verge de la Cinta, Tortosa
  - Doctor Peset University Hospital, Valencia
  - Hospital La Fe, Valencia
- University Hospital Zürich, Zurich, Switzerland
- United Kingdom (153):
  - Basildon Hospital, Basildon, England
  - Basingstoke and North Hampshire Hospital, Basingstoke, England
  - Royal United Hospital, Bath, Bath, England
  - Queen Elizabeth Hospital Birmingham, Birmingham, England
  - Birmingham City Hospital, Birmingham, England
  - Royal Blackburn Teaching Hospital, Blackburn, England
  - Pilgrim Hospital ULHT, Boston, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Royal Sussex County Hospital, Brighton, England
  - Southmead Hospital, Bristol, England
  - Bristol Royal Infirmary, Bristol, England
  - Queen's Hospital, Burton, Burton-on-Trent, England
  - Royal Papworth Hospital, Cambridge, England
  - Addenbrookes Hospital, Cambridge, England
  - North Cumberland Infirmary, Carlisle, England
  - St Peter's Hospital, Chertsey, England
  - Countess of Chester Hospital, Chester, England
  - Chesterfield Royal Hospital, Chesterfield, England
  - Colchester Hospital, Colchester, England
  - University Hospital Coventry, Coventry, England
  - Darlington Memorial Hospital, Darlington, England
  - Darent Valley Hospital, Dartford, England
  - Russells Hall Hospital, Dudley, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Frimley Park Hospital, Frimley, England
  - Queen Elizabeth Hospital Gateshead, Gateshead, England
  - Medway Maritime Hospital, Gillingham, England
  - James Paget University Hospital, Great Yarmouth, England
  - Royal Surrey County Hospital, Guildford, England
  - Northwick Park Hospital, Harrow, England
  - Hereford County Hospital, Hereford, England
  - Barnet Hospital, High Barnet, England
  - Huddersfield Royal Infirmary, Huddersfield, England
  - King George Hospital, Ilford, England
  - Ipswich Hospital, Ipswich, England
  - Kettering Hospital, Kettering, England
  - Leeds General Infirmary, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Glenfield Hospital, Leicester, England
  - Lincoln County Hospital, Lincoln, England
  - Liverpool Heart and Chest Hospital, Liverpool, England
  - Alder Hey Hospital, Liverpool, England
  - Royal Liverpool University Hospital, Liverpool, England
  - University Hospital Aintree, Liverpool, England
  - Croydon University Hospital, London, England
  - Royal London Hospital, London, England
  - Whipps Cross Hospital, London, England
  - Newham University Hospital, London, England
  - St Bartholomew's Hospital, London, England
  - North Middlesex University Hospital, London, England
  - Royal Free Hospital, London, England
  - St Thomas Hospital, London, England
  - Guy's Hospital, London, England
  - Queen Elizabeth Hospital, Woolwich, London, England
  - King's College Hospital, London, England
  - St George's University Hospital, London, England
  - Royal Marsden Hospital, London, England
  - Royal Brompton Hospital, London, England
  - Hammersmith Hospital, London, England
  - St Mary's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Luton and Dunstable University Hospital, Luton, England
  - Maidstone Hospital, Maidstone, England
  - Manchester Royal Infirmary, Manchester, England
  - The Christie Hospital, Manchester, England
  - Wythenshawe Hospital, Manchester, England
  - North Manchester General Hospital, Manchester, England
  - Arrowe Park Hospital, Metropolitan Borough of Wirral, England
  - The James Cook University Hospital, Middlesbrough, England
  - Milton Keynes University Hospital, Milton Keynes, England
  - Royal Victoria Infirmary, Newcastle, Newcastle, England
  - Newcastle Freeman Hospital, Newcastle, England
  - Northampton General Hospital, Northampton, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - City Hospital Nottingham, Nottingham, England
  - Queen's Medical Centre - Nottingham University Hospitals NHS Trust, Nottingham, England
  - George Eliot Hospital, Nuneaton, England
  - Royal Oldham Hospital, Oldham, England
  - Princess Royal University Hospital, Orpington, England
  - John Radcliffe Hospital, Oxford, England
  - Derriford Hospital, Plymouth, England
  - Poole Hospital NHS Foundation Trust, Poole, England
  - Queen Alexandra Hospital, Portsmouth, England
  - Whiston Hospital, Prescot, England
  - Royal Preston Hospital, Preston, England
  - Royal Berkshire Hospital, Reading, England
  - Alexandra Hospital, Redditch, Redditch, England
  - Queen's Hospital Romford, Romford, England
  - Rotherham Hospital, Rotherham, England
  - Tunbridge Wells Hospital - Maidstone and Tunbridge Wells NHS Trust, Royal Tunbridge Wells, England
  - Salford Royal Hospital, Salford, England
  - Salisbury District Hospital, Salisbury, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Northern General Hospital, Sheffield, England
  - Wexham Park Hospital, Slough, England
  - South Tyneside District Hospital, South Shields, England
  - Southampton General Hospital, Southampton, England
  - Stepping Hill Hospital, Stockport, England
  - University Hospital of North Tees, Stockton-on-Tees, England
  - Royal Stoke University Hospital, Stoke-on-Trent, England
  - Sunderland Royal Hospital, Sunderland, England
  - King's Mill Hospital, Sutton in Ashfield, England
  - Great Western Hospital, Swindon, England
  - Western General Hospital, Swindon, England
  - Musgrove Park Hospital, Taunton, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, England
  - Harefield Hospital, Uxbridge, England
  - Watford General Hospital, Watford, England
  - Southend Hospital, Westcliff-on-Sea, England
  - West Cumberland Hospital, Whitehaven, England
  - Royal Albert Edward Infirmary, Wigan, England
  - Royal Hampshire County Hospital, Winchester, England
  - New Cross Hospital Wolverhampton, Wolverhampton, England
  - Worcestershire Royal Hospital, Worcester, England
  - York Teaching Hospital, York, England
  - Antrim Area Hospital, Antrim, Northern Ireland
  - Royal Victoria Hospital Belfast, Belfast, Northern Ireland
  - Mater Hospital, Belfast, Northern Ireland
  - Belfast City Hospital, Belfast, Northern Ireland
  - Altnagelvin Hospital, Londonderry, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Queen Elizabeth University Hospital, Glasgow, Glasgow, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Neville Hall Hospital, Abergavenny, Wales
  - Glan Clwyd Hospital, Bodelwyddan, Wales
  - Princess of Wales Hospital, Bridgend, Wales
  - Cardiff and Vale University Hospital Wales, Cardiff, Wales
  - Glangwilli Hospital, Carmarthen, Wales
  - Grange University Hospital, Cwmbran, Wales
  - Royal Gwent Hospital, Newport, Wales
  - Royal Glamorgan Hospital, Pont-y-clun, Wales
  - Morriston Hospital, Swansea, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales
  - Ulster Hospital, Belfast
  - Bristol Royal Childrens Hospital, Bristol
  - Fairfield General Hospital, Bury
  - Leighton Hospital, Crewe
  - Dorset County Hospital, Dorchester
  - Gloucester Royal Hospital, Gloucester
  - The Princess Royal Hospital Haywards Heath, Haywards Heath
  - St. James University Hospital, Leeds
  - Homerton Hospital, London
  - University College London Hospital, London
  - Chelsea and Westminster Hospital, London
  - Queen Elizabeth and Queen Mother Hospital, Margate
  - Newcastle Royal Victoria Infirmary (Paediatrics), Newcastle upon Tyne
  - North Tyneside General Hospital, North Shields
  - Warwick Hospital, Warwick
  - Sandwell General Hospital, West Bromwich

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Derde L, Gordon AC, Mouncey PR, Al-Beidh F, Rowan KM, Nichol AD, Arabi YM, Annane D, Beane A, Beasley R, Bonten MJM, Bradbury CA, Brunkhorst FM, Buzgau A, Buxton M, Cheng AC, Cooper N, Cove M, Cremer OL, Detry MA, Duffy EJ, Estcourt LJ, Fitzgerald M, Galea J, Goossens H, Haniffa R, Hills TE, Huang DT, Ichihara N, King A, Lamontagne F, Lawler PR, Leavis HL, Lewis RJ, Litton E, Marshall JC, Mayr FB, McAuley DF, McGlothlin A, McGuinness SP, McVerry BJ, Morpeth SC, Murthy S, Netea MG, Ogungbenro K, Orr K, Parke RL, Parker JC, Patanwala AE, Pettila V, Reyes LF, Saito H, Santos MS, Saunders CT, Seymour CW, Shankar-Hari M, Sligl WI, Turgeon AF, Turner AM, Tong SYC, Vaara S, Youngstein T, Zarychanski R, Green C, Higgins AM, McArthur CJ, Berry LR, Lorenzi E, Berry S, Webb SA, Angus DC, van de Veerdonk FL. Tocilizumab, sarilumab and anakinra in critically ill patients with COVID-19: a randomised, controlled, open-label, adaptive platform trial. Thorax. 2025 Jul 15;80(8):530-539. doi: 10.1136/thorax-2024-222488. PMID 40360262
- [Derived] REMAP-CAP Investigators; Angus DC. Effect of hydrocortisone on mortality in patients with severe community-acquired pneumonia : The REMAP-CAP Corticosteroid Domain Randomized Clinical Trial. Intensive Care Med. 2025 Apr;51(4):665-680. doi: 10.1007/s00134-025-07861-w. Epub 2025 Apr 22. PMID 40261382
- [Derived] REMAP-CAP Investigators; Hills TE, Lorenzi E, Berry LR, Shyamsundar M, Al-Beidh F, Annane D, Arabi Y, Aryal D, Au C, Beane A, Bhimani Z, Bonten M, Bradbury CA, Brunkhorst FM, Burrell A, Buxton M, Calfee CS, Cecconi M, Cheng AC, Cove ME, Detry MA, Estcourt LJ, Fitzgerald M, Goligher EC, Goossens H, Green C, Haniffa R, Harrison DA, Hashmi M, Higgins AM, Horvat C, Huang DT, Ichihara N, Jayakumar D, Kruger PS, Lamontagne F, Lampro L, Lawler PR, Marshall JC, Mason AJ, McGlothlin A, McGuinness S, McQuilten ZK, McVerry BJ, Mouncey PR, Murthy S, Neal MD, Nichol AD, O'Kane CM, Parke RL, Parker JC, Rabindrarajan E, Reyes LF, Rowan KM, Saito H, Santos M, Saunders CT, Seymour CW, Shankar-Hari M, Sinha P, Thompson BT, Turgeon AF, Turner AM, van de Veerdonk F, Weis S, Young IS, Zarychanski R, Lewis RJ, McArthur CJ, Angus DC, Berry SM, Derde LPG, Webb SA, Gordon AC, McAuley DF. Simvastatin in Critically Ill Patients with Covid-19. N Engl J Med. 2023 Dec 21;389(25):2341-2354. doi: 10.1056/NEJMoa2309995. Epub 2023 Oct 25. PMID 37888913
- [Derived] LOVIT-COVID Investigators, on behalf of the Canadian Critical Care Trials Group, and the REMAP-CAP Investigators; Adhikari NKJ, Hashmi M, Tirupakuzhi Vijayaraghavan BK, Haniffa R, Beane A, Webb SA, Angus DC, Gordon AC, Cook DJ, Guyatt GH, Berry LR, Lorenzi E, Mouncey PR, Au C, Pinto R, Menard J, Sprague S, Masse MH, Huang DT, Heyland DK, Nichol AD, McArthur CJ, de Man A, Al-Beidh F, Annane D, Anstey M, Arabi YM, Battista MC, Berry S, Bhimani Z, Bonten MJM, Bradbury CA, Brant EB, Brunkhorst FM, Burrell A, Buxton M, Cecconi M, Cheng AC, Cohen D, Cove ME, Day AG, Derde LPG, Detry MA, Estcourt LJ, Fagbodun EO, Fitzgerald M, Goossens H, Green C, Higgins AM, Hills TE, Horvat C, Ichihara N, Jayakumar D, Kanji S, Khoso MN, Lawler PR, Lewis RJ, Litton E, Marshall JC, McAuley DF, McGlothlin A, McGuinness SP, McQuilten ZK, McVerry BJ, Murthy S, Parke RL, Parker JC, Reyes LF, Rowan KM, Saito H, Salahuddin N, Santos MS, Saunders CT, Seymour CW, Shankar-Hari M, Tolppa T, Trapani T, Turgeon AF, Turner AM, Udy AA, van de Veerdonk FL, Zarychanski R, Lamontagne F. Intravenous Vitamin C for Patients Hospitalized With COVID-19: Two Harmonized Randomized Clinical Trials. JAMA. 2023 Nov 14;330(18):1745-1759. doi: 10.1001/jama.2023.21407. PMID 37877585
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818
- [Derived] Writing Committee for the REMAP-CAP Investigators; Lawler PR, Derde LPG, van de Veerdonk FL, McVerry BJ, Huang DT, Berry LR, Lorenzi E, van Kimmenade R, Gommans F, Vaduganathan M, Leaf DE, Baron RM, Kim EY, Frankfurter C, Epelman S, Kwan Y, Grieve R, O'Neill S, Sadique Z, Puskarich M, Marshall JC, Higgins AM, Mouncey PR, Rowan KM, Al-Beidh F, Annane D, Arabi YM, Au C, Beane A, van Bentum-Puijk W, Bonten MJM, Bradbury CA, Brunkhorst FM, Burrell A, Buzgau A, Buxton M, Cecconi M, Cheng AC, Cove M, Detry MA, Estcourt LJ, Ezekowitz J, Fitzgerald M, Gattas D, Godoy LC, Goossens H, Haniffa R, Harrison DA, Hills T, Horvat CM, Ichihara N, Lamontagne F, Linstrum KM, McAuley DF, McGlothlin A, McGuinness SP, McQuilten Z, Murthy S, Nichol AD, Owen DRJ, Parke RL, Parker JC, Pollock KM, Reyes LF, Saito H, Santos MS, Saunders CT, Seymour CW, Shankar-Hari M, Singh V, Turgeon AF, Turner AM, Zarychanski R, Green C, Lewis RJ, Angus DC, Berry S, Gordon AC, McArthur CJ, Webb SA. Effect of Angiotensin-Converting Enzyme Inhibitor and Angiotensin Receptor Blocker Initiation on Organ Support-Free Days in Patients Hospitalized With COVID-19: A Randomized Clinical Trial. JAMA. 2023 Apr 11;329(14):1183-1196. doi: 10.1001/jama.2023.4480. PMID 37039790
- [Derived] Nurmi V, Knight C, Estcourt L, Hepojoki J, Lamikanra AA, Tsang HP, Roberts DJ, Polack FP, Simmonds P, Hedman K, Alvarez-Paggi D, Harvala H. The Relationship Between SARS-CoV-2 Neutralizing Antibody Titers and Avidity in Plasma Collected From Convalescent Nonvaccinated and Vaccinated Blood Donors. J Infect Dis. 2023 Aug 11;228(3):245-250. doi: 10.1093/infdis/jiad070. PMID 36967714
- [Derived] Goligher EC, Lawler PR, Jensen TP, Talisa V, Berry LR, Lorenzi E, McVerry BJ, Chang CH, Leifer E, Bradbury C, Berger J, Hunt BJ, Castellucci LA, Kornblith LZ, Gordon AC, McArthur C, Webb S, Hochman J, Neal MD, Zarychanski R, Berry S, Angus DC; REMAP-CAP, ATTACC, and ACTIV-4a Investigators. Heterogeneous Treatment Effects of Therapeutic-Dose Heparin in Patients Hospitalized for COVID-19. JAMA. 2023 Apr 4;329(13):1066-1077. doi: 10.1001/jama.2023.3651. PMID 36942550
- [Derived] REMAP-CAP Writing Committee for the REMAP-CAP Investigators; Bradbury CA, Lawler PR, Stanworth SJ, McVerry BJ, McQuilten Z, Higgins AM, Mouncey PR, Al-Beidh F, Rowan KM, Berry LR, Lorenzi E, Zarychanski R, Arabi YM, Annane D, Beane A, van Bentum-Puijk W, Bhimani Z, Bihari S, Bonten MJM, Brunkhorst FM, Buzgau A, Buxton M, Carrier M, Cheng AC, Cove M, Detry MA, Estcourt LJ, Fitzgerald M, Girard TD, Goligher EC, Goossens H, Haniffa R, Hills T, Huang DT, Horvat CM, Hunt BJ, Ichihara N, Lamontagne F, Leavis HL, Linstrum KM, Litton E, Marshall JC, McAuley DF, McGlothlin A, McGuinness SP, Middeldorp S, Montgomery SK, Morpeth SC, Murthy S, Neal MD, Nichol AD, Parke RL, Parker JC, Reyes LF, Saito H, Santos MS, Saunders CT, Serpa-Neto A, Seymour CW, Shankar-Hari M, Singh V, Tolppa T, Turgeon AF, Turner AM, van de Veerdonk FL, Green C, Lewis RJ, Angus DC, McArthur CJ, Berry S, Derde LPG, Webb SA, Gordon AC. Effect of Antiplatelet Therapy on Survival and Organ Support-Free Days in Critically Ill Patients With COVID-19: A Randomized Clinical Trial. JAMA. 2022 Apr 5;327(13):1247-1259. doi: 10.1001/jama.2022.2910. PMID 35315874
- [Derived] Writing Committee for the REMAP-CAP Investigators; Estcourt LJ, Turgeon AF, McQuilten ZK, McVerry BJ, Al-Beidh F, Annane D, Arabi YM, Arnold DM, Beane A, Begin P, van Bentum-Puijk W, Berry LR, Bhimani Z, Birchall JE, Bonten MJM, Bradbury CA, Brunkhorst FM, Buxton M, Callum JL, Chasse M, Cheng AC, Cove ME, Daly J, Derde L, Detry MA, De Jong M, Evans A, Fergusson DA, Fish M, Fitzgerald M, Foley C, Goossens H, Gordon AC, Gosbell IB, Green C, Haniffa R, Harvala H, Higgins AM, Hills TE, Hoad VC, Horvat C, Huang DT, Hudson CL, Ichihara N, Laing E, Lamikanra AA, Lamontagne F, Lawler PR, Linstrum K, Litton E, Lorenzi E, MacLennan S, Marshall J, McAuley DF, McDyer JF, McGlothlin A, McGuinness S, Miflin G, Montgomery S, Mouncey PR, Murthy S, Nichol A, Parke R, Parker JC, Priddee N, Purcell DFJ, Reyes LF, Richardson P, Robitaille N, Rowan KM, Rynne J, Saito H, Santos M, Saunders CT, Serpa Neto A, Seymour CW, Silversides JA, Tinmouth AA, Triulzi DJ, Turner AM, van de Veerdonk F, Walsh TS, Wood EM, Berry S, Lewis RJ, Menon DK, McArthur C, Zarychanski R, Angus DC, Webb SA, Roberts DJ, Shankar-Hari M. Effect of Convalescent Plasma on Organ Support-Free Days in Critically Ill Patients With COVID-19: A Randomized Clinical Trial. JAMA. 2021 Nov 2;326(17):1690-1702. doi: 10.1001/jama.2021.18178. PMID 34606578
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] REMAP-CAP Investigators; ACTIV-4a Investigators; ATTACC Investigators; Goligher EC, Bradbury CA, McVerry BJ, Lawler PR, Berger JS, Gong MN, Carrier M, Reynolds HR, Kumar A, Turgeon AF, Kornblith LZ, Kahn SR, Marshall JC, Kim KS, Houston BL, Derde LPG, Cushman M, Tritschler T, Angus DC, Godoy LC, McQuilten Z, Kirwan BA, Farkouh ME, Brooks MM, Lewis RJ, Berry LR, Lorenzi E, Gordon AC, Ahuja T, Al-Beidh F, Annane D, Arabi YM, Aryal D, Baumann Kreuziger L, Beane A, Bhimani Z, Bihari S, Billett HH, Bond L, Bonten M, Brunkhorst F, Buxton M, Buzgau A, Castellucci LA, Chekuri S, Chen JT, Cheng AC, Chkhikvadze T, Coiffard B, Contreras A, Costantini TW, de Brouwer S, Detry MA, Duggal A, Dzavik V, Effron MB, Eng HF, Escobedo J, Estcourt LJ, Everett BM, Fergusson DA, Fitzgerald M, Fowler RA, Froess JD, Fu Z, Galanaud JP, Galen BT, Gandotra S, Girard TD, Goodman AL, Goossens H, Green C, Greenstein YY, Gross PL, Haniffa R, Hegde SM, Hendrickson CM, Higgins AM, Hindenburg AA, Hope AA, Horowitz JM, Horvat CM, Huang DT, Hudock K, Hunt BJ, Husain M, Hyzy RC, Jacobson JR, Jayakumar D, Keller NM, Khan A, Kim Y, Kindzelski A, King AJ, Knudson MM, Kornblith AE, Kutcher ME, Laffan MA, Lamontagne F, Le Gal G, Leeper CM, Leifer ES, Lim G, Gallego Lima F, Linstrum K, Litton E, Lopez-Sendon J, Lother SA, Marten N, Saud Marinez A, Martinez M, Mateos Garcia E, Mavromichalis S, McAuley DF, McDonald EG, McGlothlin A, McGuinness SP, Middeldorp S, Montgomery SK, Mouncey PR, Murthy S, Nair GB, Nair R, Nichol AD, Nicolau JC, Nunez-Garcia B, Park JJ, Park PK, Parke RL, Parker JC, Parnia S, Paul JD, Pompilio M, Quigley JG, Rosenson RS, Rost NS, Rowan K, Santos FO, Santos M, Santos MO, Satterwhite L, Saunders CT, Schreiber J, Schutgens REG, Seymour CW, Siegal DM, Silva DG Jr, Singhal AB, Slutsky AS, Solvason D, Stanworth SJ, Turner AM, van Bentum-Puijk W, van de Veerdonk FL, van Diepen S, Vazquez-Grande G, Wahid L, Wareham V, Widmer RJ, Wilson JG, Yuriditsky E, Zhong Y, Berry SM, McArthur CJ, Neal MD, Hochman JS, Webb SA, Zarychanski R. Therapeutic Anticoagulation with Heparin in Critically Ill Patients with Covid-19. N Engl J Med. 2021 Aug 26;385(9):777-789. doi: 10.1056/NEJMoa2103417. Epub 2021 Aug 4. PMID 34351722
- [Derived] ATTACC Investigators; ACTIV-4a Investigators; REMAP-CAP Investigators; Lawler PR, Goligher EC, Berger JS, Neal MD, McVerry BJ, Nicolau JC, Gong MN, Carrier M, Rosenson RS, Reynolds HR, Turgeon AF, Escobedo J, Huang DT, Bradbury CA, Houston BL, Kornblith LZ, Kumar A, Kahn SR, Cushman M, McQuilten Z, Slutsky AS, Kim KS, Gordon AC, Kirwan BA, Brooks MM, Higgins AM, Lewis RJ, Lorenzi E, Berry SM, Berry LR, Aday AW, Al-Beidh F, Annane D, Arabi YM, Aryal D, Baumann Kreuziger L, Beane A, Bhimani Z, Bihari S, Billett HH, Bond L, Bonten M, Brunkhorst F, Buxton M, Buzgau A, Castellucci LA, Chekuri S, Chen JT, Cheng AC, Chkhikvadze T, Coiffard B, Costantini TW, de Brouwer S, Derde LPG, Detry MA, Duggal A, Dzavik V, Effron MB, Estcourt LJ, Everett BM, Fergusson DA, Fitzgerald M, Fowler RA, Galanaud JP, Galen BT, Gandotra S, Garcia-Madrona S, Girard TD, Godoy LC, Goodman AL, Goossens H, Green C, Greenstein YY, Gross PL, Hamburg NM, Haniffa R, Hanna G, Hanna N, Hegde SM, Hendrickson CM, Hite RD, Hindenburg AA, Hope AA, Horowitz JM, Horvat CM, Hudock K, Hunt BJ, Husain M, Hyzy RC, Iyer VN, Jacobson JR, Jayakumar D, Keller NM, Khan A, Kim Y, Kindzelski AL, King AJ, Knudson MM, Kornblith AE, Krishnan V, Kutcher ME, Laffan MA, Lamontagne F, Le Gal G, Leeper CM, Leifer ES, Lim G, Lima FG, Linstrum K, Litton E, Lopez-Sendon J, Lopez-Sendon Moreno JL, Lother SA, Malhotra S, Marcos M, Saud Marinez A, Marshall JC, Marten N, Matthay MA, McAuley DF, McDonald EG, McGlothlin A, McGuinness SP, Middeldorp S, Montgomery SK, Moore SC, Morillo Guerrero R, Mouncey PR, Murthy S, Nair GB, Nair R, Nichol AD, Nunez-Garcia B, Pandey A, Park PK, Parke RL, Parker JC, Parnia S, Paul JD, Perez Gonzalez YS, Pompilio M, Prekker ME, Quigley JG, Rost NS, Rowan K, Santos FO, Santos M, Olombrada Santos M, Satterwhite L, Saunders CT, Schutgens REG, Seymour CW, Siegal DM, Silva DG Jr, Shankar-Hari M, Sheehan JP, Singhal AB, Solvason D, Stanworth SJ, Tritschler T, Turner AM, van Bentum-Puijk W, van de Veerdonk FL, van Diepen S, Vazquez-Grande G, Wahid L, Wareham V, Wells BJ, Widmer RJ, Wilson JG, Yuriditsky E, Zampieri FG, Angus DC, McArthur CJ, Webb SA, Farkouh ME, Hochman JS, Zarychanski R. Therapeutic Anticoagulation with Heparin in Noncritically Ill Patients with Covid-19. N Engl J Med. 2021 Aug 26;385(9):790-802. doi: 10.1056/NEJMoa2105911. Epub 2021 Aug 4. PMID 34351721
- [Derived] Arabi YM, Gordon AC, Derde LPG, Nichol AD, Murthy S, Beidh FA, Annane D, Swaidan LA, Beane A, Beasley R, Berry LR, Bhimani Z, Bonten MJM, Bradbury CA, Brunkhorst FM, Buxton M, Buzgau A, Cheng A, De Jong M, Detry MA, Duffy EJ, Estcourt LJ, Fitzgerald M, Fowler R, Girard TD, Goligher EC, Goossens H, Haniffa R, Higgins AM, Hills TE, Horvat CM, Huang DT, King AJ, Lamontagne F, Lawler PR, Lewis R, Linstrum K, Litton E, Lorenzi E, Malakouti S, McAuley DF, McGlothlin A, Mcguinness S, McVerry BJ, Montgomery SK, Morpeth SC, Mouncey PR, Orr K, Parke R, Parker JC, Patanwala AE, Rowan KM, Santos MS, Saunders CT, Seymour CW, Shankar-Hari M, Tong SYC, Turgeon AF, Turner AM, Van de Veerdonk FL, Zarychanski R, Green C, Berry S, Marshall JC, McArthur C, Angus DC, Webb SA; REMAP-CAP Investigators. Lopinavir-ritonavir and hydroxychloroquine for critically ill patients with COVID-19: REMAP-CAP randomized controlled trial. Intensive Care Med. 2021 Aug;47(8):867-886. doi: 10.1007/s00134-021-06448-5. Epub 2021 Jul 12. PMID 34251506
- [Derived] REMAP-CAP Investigators; Gordon AC, Mouncey PR, Al-Beidh F, Rowan KM, Nichol AD, Arabi YM, Annane D, Beane A, van Bentum-Puijk W, Berry LR, Bhimani Z, Bonten MJM, Bradbury CA, Brunkhorst FM, Buzgau A, Cheng AC, Detry MA, Duffy EJ, Estcourt LJ, Fitzgerald M, Goossens H, Haniffa R, Higgins AM, Hills TE, Horvat CM, Lamontagne F, Lawler PR, Leavis HL, Linstrum KM, Litton E, Lorenzi E, Marshall JC, Mayr FB, McAuley DF, McGlothlin A, McGuinness SP, McVerry BJ, Montgomery SK, Morpeth SC, Murthy S, Orr K, Parke RL, Parker JC, Patanwala AE, Pettila V, Rademaker E, Santos MS, Saunders CT, Seymour CW, Shankar-Hari M, Sligl WI, Turgeon AF, Turner AM, van de Veerdonk FL, Zarychanski R, Green C, Lewis RJ, Angus DC, McArthur CJ, Berry S, Webb SA, Derde LPG. Interleukin-6 Receptor Antagonists in Critically Ill Patients with Covid-19. N Engl J Med. 2021 Apr 22;384(16):1491-1502. doi: 10.1056/NEJMoa2100433. Epub 2021 Feb 25. PMID 33631065
- [Derived] UPMC REMAP-COVID Group, on behalf of the REMAP-CAP Investigators. Implementation of the Randomized Embedded Multifactorial Adaptive Platform for COVID-19 (REMAP-COVID) trial in a US health system-lessons learned and recommendations. Trials. 2021 Jan 28;22(1):100. doi: 10.1186/s13063-020-04997-6. PMID 33509275
- [Derived] Tume LN, Menzies JC, Ray S, Scholefield BR; UK Paediatric Intensive Care Society Study Group. Research Priorities for U.K. Pediatric Critical Care in 2019: Healthcare Professionals' and Parents' Perspectives. Pediatr Crit Care Med. 2021 May 1;22(5):e294-e301. doi: 10.1097/PCC.0000000000002647. PMID 33394942
- [Derived] Angus DC, Derde L, Al-Beidh F, Annane D, Arabi Y, Beane A, van Bentum-Puijk W, Berry L, Bhimani Z, Bonten M, Bradbury C, Brunkhorst F, Buxton M, Buzgau A, Cheng AC, de Jong M, Detry M, Estcourt L, Fitzgerald M, Goossens H, Green C, Haniffa R, Higgins AM, Horvat C, Hullegie SJ, Kruger P, Lamontagne F, Lawler PR, Linstrum K, Litton E, Lorenzi E, Marshall J, McAuley D, McGlothin A, McGuinness S, McVerry B, Montgomery S, Mouncey P, Murthy S, Nichol A, Parke R, Parker J, Rowan K, Sanil A, Santos M, Saunders C, Seymour C, Turner A, van de Veerdonk F, Venkatesh B, Zarychanski R, Berry S, Lewis RJ, McArthur C, Webb SA, Gordon AC; Writing Committee for the REMAP-CAP Investigators; Al-Beidh F, Angus D, Annane D, Arabi Y, van Bentum-Puijk W, Berry S, Beane A, Bhimani Z, Bonten M, Bradbury C, Brunkhorst F, Buxton M, Cheng A, De Jong M, Derde L, Estcourt L, Goossens H, Gordon A, Green C, Haniffa R, Lamontagne F, Lawler P, Litton E, Marshall J, McArthur C, McAuley D, McGuinness S, McVerry B, Montgomery S, Mouncey P, Murthy S, Nichol A, Parke R, Rowan K, Seymour C, Turner A, van de Veerdonk F, Webb S, Zarychanski R, Campbell L, Forbes A, Gattas D, Heritier S, Higgins L, Kruger P, Peake S, Presneill J, Seppelt I, Trapani T, Young P, Bagshaw S, Daneman N, Ferguson N, Misak C, Santos M, Hullegie S, Pletz M, Rohde G, Rowan K, Alexander B, Basile K, Girard T, Horvat C, Huang D, Linstrum K, Vates J, Beasley R, Fowler R, McGloughlin S, Morpeth S, Paterson D, Venkatesh B, Uyeki T, Baillie K, Duffy E, Fowler R, Hills T, Orr K, Patanwala A, Tong S, Netea M, Bihari S, Carrier M, Fergusson D, Goligher E, Haidar G, Hunt B, Kumar A, Laffan M, Lawless P, Lother S, McCallum P, Middeldopr S, McQuilten Z, Neal M, Pasi J, Schutgens R, Stanworth S, Turgeon A, Weissman A, Adhikari N, Anstey M, Brant E, de Man A, Lamonagne F, Masse MH, Udy A, Arnold D, Begin P, Charlewood R, Chasse M, Coyne M, Cooper J, Daly J, Gosbell I, Harvala-Simmonds H, Hills T, MacLennan S, Menon D, McDyer J, Pridee N, Roberts D, Shankar-Hari M, Thomas H, Tinmouth A, Triulzi D, Walsh T, Wood E, Calfee C, O'Kane C, Shyamsundar M, Sinha P, Thompson T, Young I, Bihari S, Hodgson C, Laffey J, McAuley D, Orford N, Neto A, Detry M, Fitzgerald M, Lewis R, McGlothlin A, Sanil A, Saunders C, Berry L, Lorenzi E, Miller E, Singh V, Zammit C, van Bentum Puijk W, Bouwman W, Mangindaan Y, Parker L, Peters S, Rietveld I, Raymakers K, Ganpat R, Brillinger N, Markgraf R, Ainscough K, Brickell K, Anjum A, Lane JB, Richards-Belle A, Saull M, Wiley D, Bion J, Connor J, Gates S, Manax V, van der Poll T, Reynolds J, van Beurden M, Effelaar E, Schotsman J, Boyd C, Harland C, Shearer A, Wren J, Clermont G, Garrard W, Kalchthaler K, King A, Ricketts D, Malakoutis S, Marroquin O, Music E, Quinn K, Cate H, Pearson K, Collins J, Hanson J, Williams P, Jackson S, Asghar A, Dyas S, Sutu M, Murphy S, Williamson D, Mguni N, Potter A, Porter D, Goodwin J, Rook C, Harrison S, Williams H, Campbell H, Lomme K, Williamson J, Sheffield J, van't Hoff W, McCracken P, Young M, Board J, Mart E, Knott C, Smith J, Boschert C, Affleck J, Ramanan M, D'Souza R, Pateman K, Shakih A, Cheung W, Kol M, Wong H, Shah A, Wagh A, Simpson J, Duke G, Chan P, Cartner B, Hunter S, Laver R, Shrestha T, Regli A, Pellicano A, McCullough J, Tallott M, Kumar N, Panwar R, Brinkerhoff G, Koppen C, Cazzola F, Brain M, Mineall S, Fischer R, Biradar V, Soar N, White H, Estensen K, Morrison L, Smith J, Cooper M, Health M, Shehabi Y, Al-Bassam W, Hulley A, Whitehead C, Lowrey J, Gresha R, Walsham J, Meyer J, Harward M, Venz E, Williams P, Kurenda C, Smith K, Smith M, Garcia R, Barge D, Byrne D, Byrne K, Driscoll A, Fortune L, Janin P, Yarad E, Hammond N, Bass F, Ashelford A, Waterson S, Wedd S, McNamara R, Buhr H, Coles J, Schweikert S, Wibrow B, Rauniyar R, Myers E, Fysh E, Dawda A, Mevavala B, Litton E, Ferrier J, Nair P, Buscher H, Reynolds C, Santamaria J, Barbazza L, Homes J, Smith R, Murray L, Brailsford J, Forbes L, Maguire T, Mariappa V, Smith J, Simpson S, Maiden M, Bone A, Horton M, Salerno T, Sterba M, Geng W, Depuydt P, De Waele J, De Bus L, Fierens J, Bracke S, Reeve B, Dechert W, Chasse M, Carrier FM, Boumahni D, Benettaib F, Ghamraoui A, Bellemare D, Cloutier E, Francoeur C, Lamontagne F, D'Aragon F, Carbonneau E, Leblond J, Vazquez-Grande G, Marten N, Wilson M, Albert M, Serri K, Cavayas A, Duplaix M, Williams V, Rochwerg B, Karachi T, Oczkowski S, Centofanti J, Millen T, Duan E, Tsang J, Patterson L, English S, Watpool I, Porteous R, Miezitis S, McIntyre L, Brochard L, Burns K, Sandhu G, Khalid I, Binnie A, Powell E, McMillan A, Luk T, Aref N, Andric Z, Cviljevic S, Dimoti R, Zapalac M, Mirkovic G, Barsic B, Kutlesa M, Kotarski V, Vujaklija Brajkovic A, Babel J, Sever H, Dragija L, Kusan I, Vaara S, Pettila L, Heinonen J, Kuitunen A, Karlsson S, Vahtera A, Kiiski H, Ristimaki S, Azaiz A, Charron C, Godement M, Geri G, Vieillard-Baron A, Pourcine F, Monchi M, Luis D, Mercier R, Sagnier A, Verrier N, Caplin C, Siami S, Aparicio C, Vautier S, Jeblaoui A, Fartoukh M, Courtin L, Labbe V, Leparco C, Muller G, Nay MA, Kamel T, Benzekri D, Jacquier S, Mercier E, Chartier D, Salmon C, Dequin P, Schneider F, Morel G, L'Hotellier S, Badie J, Berdaguer FD, Malfroy S, Mezher C, Bourgoin C, Megarbane B, Voicu S, Deye N, Malissin I, Sutterlin L, Guitton C, Darreau C, Landais M, Chudeau N, Robert A, Moine P, Heming N, Maxime V, Bossard I, Nicholier TB, Colin G, Zinzoni V, Maquigneau N, Finn A, Kress G, Hoff U, Friedrich Hinrichs C, Nee J, Pletz M, Hagel S, Ankert J, Kolanos S, Bloos F, Petros S, Pasieka B, Kunz K, Appelt P, Schutze B, Kluge S, Nierhaus A, Jarczak D, Roedl K, Weismann D, Frey A, Klinikum Neukolln V, Reill L, Distler M, Maselli A, Belteczki J, Magyar I, Fazekas A, Kovacs S, Szoke V, Szigligeti G, Leszkoven J, Collins D, Breen P, Frohlich S, Whelan R, McNicholas B, Scully M, Casey S, Kernan M, Doran P, O'Dywer M, Smyth M, Hayes L, Hoiting O, Peters M, Rengers E, Evers M, Prinssen A, Bosch Ziekenhuis J, Simons K, Rozendaal W, Polderman F, de Jager P, Moviat M, Paling A, Salet A, Rademaker E, Peters AL, de Jonge E, Wigbers J, Guilder E, Butler M, Cowdrey KA, Newby L, Chen Y, Simmonds C, McConnochie R, Ritzema Carter J, Henderson S, Van Der Heyden K, Mehrtens J, Williams T, Kazemi A, Song R, Lai V, Girijadevi D, Everitt R, Russell R, Hacking D, Buehner U, Williams E, Browne T, Grimwade K, Goodson J, Keet O, Callender O, Martynoga R, Trask K, Butler A, Schischka L, Young C, Lesona E, Olatunji S, Robertson Y, Jose N, Amaro dos Santos Catorze T, de Lima Pereira TNA, Neves Pessoa LM, Castro Ferreira RM, Pereira Sousa Bastos JM, Aysel Florescu S, Stanciu D, Zaharia MF, Kosa AG, Codreanu D, Marabi Y, Al Qasim E, Moneer Hagazy M, Al Swaidan L, Arishi H, Munoz-Bermudez R, Marin-Corral J, Salazar Degracia A, Parrilla Gomez F, Mateo Lopez MI, Rodriguez Fernandez J, Carcel Fernandez S, Carmona Flores R, Leon Lopez R, de la Fuente Martos C, Allan A, Polgarova P, Farahi N, McWilliam S, Hawcutt D, Rad L, O'Malley L, Whitbread J, Kelsall O, Wild L, Thrush J, Wood H, Austin K, Donnelly A, Kelly M, O'Kane S, McClintock D, Warnock M, Johnston P, Gallagher LJ, Mc Goldrick C, Mc Master M, Strzelecka A, Jha R, Kalogirou M, Ellis C, Krishnamurthy V, Deelchand V, Silversides J, McGuigan P, Ward K, O'Neill A, Finn S, Phillips B, Mullan D, Oritz-Ruiz de Gordoa L, Thomas M, Sweet K, Grimmer L, Johnson R, Pinnell J, Robinson M, Gledhill L, Wood T, Morgan M, Cole J, Hill H, Davies M, Antcliffe D, Templeton M, Rojo R, Coghlan P, Smee J, Mackay E, Cort J, Whileman A, Spencer T, Spittle N, Kasipandian V, Patel A, Allibone S, Genetu RM, Ramali M, Ghosh A, Bamford P, London E, Cawley K, Faulkner M, Jeffrey H, Smith T, Brewer C, Gregory J, Limb J, Cowton A, O'Brien J, Nikitas N, Wells C, Lankester L, Pulletz M, Williams P, Birch J, Wiseman S, Horton S, Alegria A, Turki S, Elsefi T, Crisp N, Allen L, McCullagh I, Robinson P, Hays C, Babio-Galan M, Stevenson H, Khare D, Pinder M, Selvamoni S, Gopinath A, Pugh R, Menzies D, Mackay C, Allan E, Davies G, Puxty K, McCue C, Cathcart S, Hickey N, Ireland J, Yusuff H, Isgro G, Brightling C, Bourne M, Craner M, Watters M, Prout R, Davies L, Pegler S, Kyeremeh L, Arbane G, Wilson K, Gomm L, Francia F, Brett S, Sousa Arias S, Elin Hall R, Budd J, Small C, Birch J, Collins E, Henning J, Bonner S, Hugill K, Cirstea E, Wilkinson D, Karlikowski M, Sutherland H, Wilhelmsen E, Woods J, North J, Sundaran D, Hollos L, Coburn S, Walsh J, Turns M, Hopkins P, Smith J, Noble H, Depante MT, Clarey E, Laha S, Verlander M, Williams A, Huckle A, Hall A, Cooke J, Gardiner-Hill C, Maloney C, Qureshi H, Flint N, Nicholson S, Southin S, Nicholson A, Borgatta B, Turner-Bone I, Reddy A, Wilding L, Chamara Warnapura L, Agno Sathianathan R, Golden D, Hart C, Jones J, Bannard-Smith J, Henry J, Birchall K, Pomeroy F, Quayle R, Makowski A, Misztal B, Ahmed I, KyereDiabour T, Naiker K, Stewart R, Mwaura E, Mew L, Wren L, Willams F, Innes R, Doble P, Hutter J, Shovelton C, Plumb B, Szakmany T, Hamlyn V, Hawkins N, Lewis S, Dell A, Gopal S, Ganguly S, Smallwood A, Harris N, Metherell S, Lazaro JM, Newman T, Fletcher S, Nortje J, Fottrell-Gould D, Randell G, Zaman M, Elmahi E, Jones A, Hall K, Mills G, Ryalls K, Bowler H, Sall J, Bourne R, Borrill Z, Duncan T, Lamb T, Shaw J, Fox C, Moreno Cuesta J, Xavier K, Purohit D, Elhassan M, Bakthavatsalam D, Rowland M, Hutton P, Bashyal A, Davidson N, Hird C, Chhablani M, Phalod G, Kirkby A, Archer S, Netherton K, Reschreiter H, Camsooksai J, Patch S, Jenkins S, Pogson D, Rose S, Daly Z, Brimfield L, Claridge H, Parekh D, Bergin C, Bates M, Dasgin J, McGhee C, Sim M, Hay SK, Henderson S, Phull MK, Zaidi A, Pogreban T, Rosaroso LP, Harvey D, Lowe B, Meredith M, Ryan L, Hormis A, Walker R, Collier D, Kimpton S, Oakley S, Rooney K, Rodden N, Hughes E, Thomson N, McGlynn D, Walden A, Jacques N, Coles H, Tilney E, Vowell E, Schuster-Bruce M, Pitts S, Miln R, Purandare L, Vamplew L, Spivey M, Bean S, Burt K, Moore L, Day C, Gibson C, Gordon E, Zitter L, Keenan S, Baker E, Cherian S, Cutler S, Roynon-Reed A, Harrington K, Raithatha A, Bauchmuller K, Ahmad N, Grecu I, Trodd D, Martin J, Wrey Brown C, Arias AM, Craven T, Hope D, Singleton J, Clark S, Rae N, Welters I, Hamilton DO, Williams K, Waugh V, Shaw D, Puthucheary Z, Martin T, Santos F, Uddin R, Somerville A, Tatham KC, Jhanji S, Black E, Dela Rosa A, Howle R, Tully R, Drummond A, Dearden J, Philbin J, Munt S, Vuylsteke A, Chan C, Victor S, Matsa R, Gellamucho M, Creagh-Brown B, Tooley J, Montague L, De Beaux F, Bullman L, Kersiake I, Demetriou C, Mitchard S, Ramos L, White K, Donnison P, Johns M, Casey R, Mattocks L, Salisbury S, Dark P, Claxton A, McLachlan D, Slevin K, Lee S, Hulme J, Joseph S, Kinney F, Senya HJ, Oborska A, Kayani A, Hadebe B, Orath Prabakaran R, Nichols L, Thomas M, Worner R, Faulkner B, Gendall E, Hayes K, Hamilton-Davies C, Chan C, Mfuko C, Abbass H, Mandadapu V, Leaver S, Forton D, Patel K, Paramasivam E, Powell M, Gould R, Wilby E, Howcroft C, Banach D, Fernandez de Pinedo Artaraz Z, Cabreros L, White I, Croft M, Holland N, Pereira R, Zaki A, Johnson D, Jackson M, Garrard H, Juhaz V, Roy A, Rostron A, Woods L, Cornell S, Pillai S, Harford R, Rees T, Ivatt H, Sundara Raman A, Davey M, Lee K, Barber R, Chablani M, Brohi F, Jagannathan V, Clark M, Purvis S, Wetherill B, Dushianthan A, Cusack R, de Courcy-Golder K, Smith S, Jackson S, Attwood B, Parsons P, Page V, Zhao XB, Oza D, Rhodes J, Anderson T, Morris S, Xia Le Tai C, Thomas A, Keen A, Digby S, Cowley N, Wild L, Southern D, Reddy H, Campbell A, Watkins C, Smuts S, Touma O, Barnes N, Alexander P, Felton T, Ferguson S, Sellers K, Bradley-Potts J, Yates D, Birkinshaw I, Kell K, Marshall N, Carr-Knott L, Summers C. Effect of Hydrocortisone on Mortality and Organ Support in Patients With Severe COVID-19: The REMAP-CAP COVID-19 Corticosteroid Domain Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1317-1329. doi: 10.1001/jama.2020.17022. PMID 32876697
- [Derived] Angus DC, Berry S, Lewis RJ, Al-Beidh F, Arabi Y, van Bentum-Puijk W, Bhimani Z, Bonten M, Broglio K, Brunkhorst F, Cheng AC, Chiche JD, De Jong M, Detry M, Goossens H, Gordon A, Green C, Higgins AM, Hullegie SJ, Kruger P, Lamontagne F, Litton E, Marshall J, McGlothlin A, McGuinness S, Mouncey P, Murthy S, Nichol A, O'Neill GK, Parke R, Parker J, Rohde G, Rowan K, Turner A, Young P, Derde L, McArthur C, Webb SA. The REMAP-CAP (Randomized Embedded Multifactorial Adaptive Platform for Community-acquired Pneumonia) Study. Rationale and Design. Ann Am Thorac Soc. 2020 Jul;17(7):879-891. doi: 10.1513/AnnalsATS.202003-192SD. PMID 32267771
- See also: global REMAP-CAP Study Website — https://www.remapcap.org/
- See also: EU REMAP-CAP Study Website — https://www.remapcap.eu/